CLINICAL TRIAL: NCT00127335
Title: Double Blind, Prospective Randomized, Crossover Study of Patients With Muscle Complaints on Statin Therapy
Brief Title: Is Myopathy Part of Statin Therapy (IMPOSTER-16)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: M-05-001 (MER004241)
Record Dates: First submitted 2005-08-04; First posted 2005-08-05 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Myopathic Conditions
Keywords: rhabdomyolysis,; myositis,; myopathy,; statin side effects,; fatty acid oxidation; Statin induced Muscle toxicity
MeSH Terms: conditions — Muscular Diseases; Rhabdomyolysis; Myositis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator)
  Interventions: Drug: cellulose placebo vs. atorvastatin
- 2 (Active Comparator): statin administration
  Interventions: Drug: cellulose placebo vs. atorvastatin

INTERVENTIONS:
Drug: cellulose placebo vs. atorvastatin — drug
  Other Names: atorvastatin

SUMMARY:
There is a significant proportion of patients complaining of muscle symptoms while on statin therapy who have a measurable difference in muscle strength or endurance and whose muscle biopsies are diagnostic for myopathy.

DETAILED DESCRIPTION:
This is a double-blinded, randomized, placebo-controlled, crossover trial. Sixty patients who are identified by their physician as having muscle pain or weakness while on statin therapy and in whom creatine kinase (CK) enzyme determinations have been normal will be enrolled voluntarily. All patients will have a percutaneous muscle biopsy prior to enrollment into the trial. These patients will be randomized in a blinded crossover fashion to either standardized statin therapy or placebo in eight week intervals. After eight weeks of drug or placebo the patients will be assessed for signs and symptoms of muscle weakness by:

* Dynamometry of grip and hip strength
* An exercise test with exhaled gas analysis
* Blood tests for cholesterol, creatine kinase, lactate
* Urine tests for organic acids

Following the first eight-week study and testing period, each patient will serve as their own control and they will enter a second eight-week study period. During the second phase they will take the opposite therapy, either drug or placebo, which they have not yet received. Sub-studies will include ten controls who have never previously received statins and ten subjects who have suffered statin-induced rhabdomyolysis. Subjects in these sub-studies will not be exposed to statin therapy and will only undergo limited testing.

ELIGIBILITY:
Inclusion Criteria:

* Primary doctor's permission
* Patient understands nature of study and has signed consent
* Patient is >21 years of age
* Patient willing to stop statin for up to 12 weeks and remain off CoQ10 for study duration
* Patient able to perform the strength and functional tests required
* Patient complains of muscle weakness or aching which he/she or his/her physician feels may be attributable to statin therapy
* CK < 350 IU
* Thyroid stimulating hormone (TSH) must be normal
* Fasting respiratory exchange ratio (RER) > 0.80 off statin for at least 4 weeks

Exclusion Criteria:

* Severe underlying illness including: Cr > 3.0, liver failure, unstable angina, symptomatic valvular heart disease, congestive heart failure, or prior cerebrovascular accident (CVA) preventing exercise testing.
* History of muscle damage (CK > 350 IU) on statins
* Underlying musculoskeletal disorder preventing muscle testing
* History of severe depression
* Taking doses of other medicines with statin sufficient to cause myopathy including: cyclosporine, erythromycin or other macrolide antibiotics; fluconazole; niacin; fibrates; or > 16 oz. of grapefruit juice daily.
* Diabetes requiring other than diet therapy
* Use of thiazolidinediones (TZD's), protease inhibitors or other drugs known to influence RER or fatty acid oxidation.
* Abnormal thyroid status
* Inability to maintain constant exercise, dietary, and drug regimen during the 16 weeks required by the study protocol.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
hip flexion | 8 weeks
oxygen consumption and anaerobic threshold | 8 weeks
muscle pathology score | at entry

SECONDARY OUTCOMES:
ability to identify blinded statin | 8 weeks
other aerobic exercise indexes | 8 weeks
fatty acid oxidation of myocyte cell cultures | at entry

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Phillips, MD, Principal Investigator — Scripps Health; Harminder Sikand, PharmD, Study Director — Scripps Mercy
Locations (1):
- Scripps Mercy Hospital, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phillips PS. Ezetimibe and statin-associated myopathy. Ann Intern Med. 2004 Oct 19;141(8):649. doi: 10.7326/0003-4819-141-8-200410190-00021. No abstract available. PMID 15492351
- [Background] Phillips PS, Phillips CT, Sullivan MJ, Naviaux RK, Haas RH. Statin myotoxicity is associated with changes in the cardiopulmonary function. Atherosclerosis. 2004 Nov;177(1):183-8. doi: 10.1016/j.atherosclerosis.2004.06.014. PMID 15488882
- [Background] Phillips PS, Haas RH, Bannykh S, Hathaway S, Gray NL, Kimura BJ, Vladutiu GD, England JD; Scripps Mercy Clinical Research Center. Statin-associated myopathy with normal creatine kinase levels. Ann Intern Med. 2002 Oct 1;137(7):581-5. doi: 10.7326/0003-4819-137-7-200210010-00009. PMID 12353945
- [Background] Antons KA, Williams CD, Baker SK, Phillips PS. Clinical perspectives of statin-induced rhabdomyolysis. Am J Med. 2006 May;119(5):400-9. doi: 10.1016/j.amjmed.2006.02.007. PMID 16651050